CLINICAL TRIAL: NCT00004941
Title: Phase III Randomized Study of Anti-Tumor Necrosis Factor Chimeric Monoclonal Antibody (cA2) for Patients With Enterocutaneous Fistulae as a Complication of Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: FDA Office of Orphan Products Development (U.S. Federal Agency)
Collaborators: Centocor, Inc. (Industry)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/13447; CENTOCOR-C0168T20; CENTOCOR-FDR001276
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2000-04

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; gastrointestinal disorders; rare disease
MeSH Terms: conditions — Crohn Disease; Gastrointestinal Diseases; Rare Diseases | interventions — Infliximab

INTERVENTIONS:
Drug: monoclonal antibody cA2

SUMMARY:
OBJECTIVES:

I. Evaluate the efficacy of chimeric monoclonal antibody (cA2) compared with placebo in closure of enterocutaneous fistulae in patients with Crohn's disease.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind, placebo controlled, multicenter study. Patients are stratified according to investigational site and number of fistulae (single vs multiple).

Patients are randomized to one of three treatment arms: Arm I: Patients receive an infusion of chimeric monoclonal antibody (cA2) on weeks 0, 2, and 6. Arm II: Patients receive an infusion of cA2 on weeks 0 and 2, and an infusion of placebo on week 6. Arm III: Patients receive an infusion of placebo on day 1 of weeks 0, 2, and 6.

Patients are followed every month for 3 months, then every 6-12 months for up to 2 years.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Crohn's disease of at least 3 months duration confirmed by radiography or endoscopy

Single or multiple draining enterocutaneous (including perianal) fistulae of at least 3 months duration

All fistulae separate and distinctly identifiable

No local complications of Crohn's disease such as strictures or abscesses

--Prior/Concurrent Therapy--

Biologic therapy:

* No prior chimeric monoclonal antibody (cA2)
* At least 3 months since treatment with other therapeutic agent targeted at reducing tumor necrosis factor (e.g., pentoxifylline or thalidomide)
* At least 4 weeks since cyclosporine

Chemotherapy:

* Concurrent methotrexate permitted if treatment began at least 3 months prior to enrollment, dose has been stable for at least 4 weeks prior to enrollment and remains stable throughout study period
* Otherwise, no methotrexate within 4 weeks prior to enrollment

Concurrent 6-mercaptopurine or azathioprine permitted if treatment began at least 6 months prior to enrollment, dose has been stable for at least 8 weeks prior to enrollment, and remains stable throughout study period Otherwise, no 6-mercaptopurine or azathioprine within 4 weeks prior to enrollment

Endocrine therapy:

* Concurrent corticosteroids (e.g., oral prednisone) permitted if dose has been stable for at least 3 weeks prior to enrollment, does not exceed 40 mg/kg, and remains stable throughout study period (dosage may be tapered after 6 weeks for some patients)
* Otherwise, no corticosteroids within 4 weeks prior to enrollment

Other:

* Concurrent antibiotics or aminosalicylates for Crohn's disease permitted if dose has been stable for at least 4 weeks prior to enrollment and remains stable throughout study period
* Otherwise, no antibiotics or aminosalicylates within 4 weeks prior to enrollment
* At least 3 months since investigational drugs

--Patient Characteristics--

Hematopoietic:

* WBC at least 3,500/mm3
* Neutrophil count at least 1,500/mm3
* Lymphocyte count at least 500/mm3
* Platelet count at least 100,000/mm3
* Hemoglobin at least 8.5 g/dL
* No severe, progressive, or uncontrolled hematologic disease

Hepatic:

* SGOT no greater than 3 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 3 times ULN
* No severe, progressive, or uncontrolled hepatic disease

Renal:

* Creatinine no greater than 1.7 mg/dL
* No severe, progressive, or uncontrolled renal disease

Cardiovascular: No severe, progressive, or uncontrolled cardiac disease

Pulmonary: No severe, progressive, or uncontrolled pulmonary disease

Neurologic: No severe, progressive, or uncontrolled neurologic or cerebral disease

Other:

* Negative pregnancy test required and no planned pregnancy within 7.5 months following first infusion
* Effective contraception required of fertile patients during and for 6 months after study
* No severe, progressive, or uncontrolled endocrine disease
* No serious infections (e.g., hepatitis, pneumonia, pyelonephritis) within prior 3 months
* No history of opportunistic infections (e.g., herpes zoster) within 2 months
* No allergy to murine proteins
* No active cytomegalovirus, Pneumocystis carinii, or drug resistant atypical mycobacterial infections
* No recent drug or alcohol abuse
* No HIV infection, ARC (AIDS-related complex) or AIDS
* Total parenteral nutrition or tube feeding not permitted
* No prior or concurrent malignancy within 5 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94
Dates: Start 1996-07; Study Completion 1996-07

CONTACTS AND LOCATIONS:
Overall Officials: Richard Vensel McCloskey, Study Chair — Centocor, Inc.